CLINICAL TRIAL: NCT02117206
Title: Protective Effects of L-arginine During Reperfusion by Femoropopliteal Bypass for Lower Limb Ischemic Syndrome in Humans
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 3262
Record Dates: First submitted 2014-03-25; First posted 2014-04-17 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-04

CONDITIONS: Skeletal Muscle Ischemia; Severe Lower Limb Ischemia; Mitochondrial Dysfunction
Keywords: L-arginine
MeSH Terms: conditions — Mitochondrial Diseases | interventions — Arginine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- L-Arginine (Active Comparator): Femoral arterial infusion of 2 g L-Arginine for 30 min
  Interventions: Drug: L-arginine (L-arginine Veyron)
- Nacl (Placebo Comparator): Femoral arterial infusion of Nacl for 30 min
  Interventions: Drug: Nacl

INTERVENTIONS:
Drug: L-arginine (L-arginine Veyron)
  Arms: L-Arginine
Drug: Nacl
  Arms: Nacl

SUMMARY:
The symptoms and severity of arterial disease is secondary to perfusion deficit. The specific alteration of the mitochondrial function of ischemic skeletal muscle plays an important role, and therapeutic enhancing mitochondrial function are associated with a clinical improvement with increase in the walking distance of the patient.

In severe ischemia, reperfusion required is accompanied by a deleterious episode through a worsening of endothelial dysfunction (impaired pathway of nitric oxide (NO)), majorant alteration of cellular energy and the hormonal and inflammatory responses. This is reperfusion syndrome, which can lead to grave consequences. Our goal is to limit mitochondrial and endothelial dysfunction (increased by the reperfusion) by stimulating the NO pathway by in situ addition of its precursor, L-arginine. Our working hypothesis is that this cellular improvement will be accompanied by an increase in systolic pressure index and an improvement in the walking distance.

Method: This is a trial with direct individual benefit, comparative, randomized, prospective, single-center, double-blind, versus placebo.

DETAILED DESCRIPTION:
2 groups of 30 patients with severe lower limb ischemia requiring femoropopliteal bypass revascularization participate in the study. The control group (placebo isoosmotic saline) will be compared to the treated group (femoral arterial infusion of 2 g L-Arginine for 30 min).

Heart rate, blood pressure and body temperature will be monitored continuously. The gastrocnemius muscle is biopsied before and 30 minutes after revascularization to analyze mitochondrial respiration and its control. Both femoral and brachial concomitant venous samples will judge the importance of muscle damage (lactate, muscle enzymes) and released mediators (cytokines, NO and endothelin) on the local and general.

Main clinical implications: L-arginine supplementation in atherosclerotic patients requiring femoropopliteal bypass to limit the initial deleterious effects of reperfusion and improve their walking distance and therefore their quality of life. Then extending this treatment to other patients with peripheral arterial disease.

ELIGIBILITY:
Inclusion Criteria:

* atherosclerotic patient with peripheral arterial disease stage 2-4 Leriche and Fontaine classification
* requiring surgical revascularization by femoropopliteal bypass
* above 18 years old

Exclusion Criteria:

* active infectious disease
* severe heart disease
* chronic renal insufficency
* pregnant women
* women of childbearing age and with no effective contraception for at least three months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-11; Primary Completion 2012-03 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Protective effect of L-Arginine on skeletal muscle: V0 and Vmax measurements ACR (Acceptor control ratio)=Vmax/V0 | Immediate post surgery muscle biopsy analysis

SECONDARY OUTCOMES:
Increase walking distance and ankle brachial index | 1 month and 3 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Fabien THAVEAU, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- SERVICE DE PHYSIOLOGIE ET D'EXPLORATIONS FONCTIONNELLES- Nouvel Hôpital Civil, HUS, Strasbourg, France